CLINICAL TRIAL: NCT01491789
Title: Virtual Sailing Simulator in Individuals With Spinal Cord Injury
Acronym: VSail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Albert Recio, M.D., Faculty, Physician, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00044093
Record Dates: First submitted 2011-12-06; First posted 2011-12-14 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; Virtual sailing; Vsail
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Virtual Sailing (Experimental): you will be doing 60 minutes of Virtual Sailing training, 1 time a week for 12 weeks
  Interventions: Device: The VSail-Access simulator

INTERVENTIONS:
Device: The VSail-Access simulator — You will be transferred to the VSail cockpit and secured. Following the trainer's instruction, you will sail the simulator around virtual courses displayed on a computer screen, using a joystick to control the rudder angle and a mainsheet to control the set of the sail. You will do this for 1 hour.
  Other Names: VSail-Access simulator

SUMMARY:
The research is being done to look at the benefits of a recreational and therapeutic program for people with spinal cord injury using the VSail-Access sailing simulator.

DETAILED DESCRIPTION:
The VSail-Access is the first sailing simulator available for people with disabilities. The VSail-Access simulator is a variation on the VSail where the cockpit is fitted with a seat. The VSail simulator is a generic sailboat cockpit powered by a pneumatic ram and custom designed software. The sailor sails the simulator around virtual courses displayed on a computer screen in the same way as a real sailboat on water. Electronic sensors provide real time feedback to match the movements of the virtual sailboat displayed on the screen with those of the simulator. Sailors can select wind strength and conditions to suit their ability.

Adults with spinal cord injury may take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, age 18-65 years, all ethnic groups.
* Spinal Cord Injury.
* Chronic injury, > 6 months from the injury.
* All ASIA neurological levels (C1-S1)
* All ASIA impairment scale A-D .
* Subjects are able to comply with procedures and follow-up.
* Subjects are medically stable, with no recent (1 month or less) inpatient admission for acute medical or surgical issues.

Exclusion Criteria:

* Cardiovascular disease as defined by previous myocardial infarction, unstable angina, requirement for anti platelet agents, congestive heart failure, or stroke NYHA Class III or IV, history of arrhythmia with hemodynamic instability.
* Uncontrolled hypertension (resting systolic BP > 160mmHg, or diastolic BP > 100mmHg consistently).
* Severe hypotension (systolic BP < 80 mmHg, or diastolic BP < 55 mmHg).
* Ventilator dependent subjects.
* Significant cognitive impairment.
* History of epileptic seizures.
* Unstable long bone fractures of the extremities.
* Subjects having Stage III or greater skin ulcerations.
* Active sailor.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Recio, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Sailing
Started | 18
Completed | 14
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Sailing
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 45 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Spinal Cord Injury Quality of Life Questionnaire (SCI QL-23
Description: This is a routine test performed for people with spinal cord injury. The SCI QL-23 is a 23-item health-related quality of life questionnaire. The subject will read the questionnaire and answer the questions; if needed ,assistance will be provided to record the answers on the form. The SCI QL-23 questionnaire will be used for all subjects.
Time Frame: Baseline
Population: Scale of 0-100, higher values represent better outcome
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Virtual Sailing
Number analyzed (Participants) | 10
score on a scale | 48.2 [0 to 100]

2. Secondary Outcome: Functional Reach Test, Level of Trunk Activation Test
Description: Two different assessments of how you are able to use your trunk will be performed. This test is performed by patient reaching forward as far as they can while seated in their wheelchair.This test will assess the activation of trunk muscle by asking the patient to perform a sit-up from the supine position
Time Frame: Baseline
Population: score on a scale of 0-30 higher values represent better outcome
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Virtual Sailing
Number analyzed (Participants) | 13
units on a scale | 13.4 [0 to 30]

3. Secondary Outcome: Grasp/Pinch Test
Description: This is a routine test performed for people with spinal cord injury. This is a standard test used to assess strength of grasp and lateral pinch. The Jamar dynamometer will be used to assess grasp and lateral pinch. This test will be performed on all subjects.
Time Frame: Baseline
Population: score on a scale from 0-200 higher values represent better outcome
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Virtual Sailing
Number analyzed (Participants) | 13
units on a scale | 55 [0 to 200]

4. Secondary Outcome: Sailing Ability Questionnaire
Description: This questionnaire will assess the subject's views about sailing, as well as the subject's perceived sailing abilities. This is a yes or no survey, Zero is no, One is yes. One means you have sailed before and zero means you have not sailed before. minimum score is 0 and maximum score is 1.
Time Frame: Baseline
Population: higher values represent better outcome
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Virtual Sailing
Number analyzed (Participants) | 13
units on a scale | 1 [0 to 1]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Virtual Sailing
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-01-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT01491789/Prot_000.pdf